CLINICAL TRIAL: NCT00336466
Title: The Erythropoietin NeuroProtective Effect: Assessment in CABG Surgery (TENPEAKS): A Randomized, Double-Blind, Placebo Controlled Proof-of-Concept Clinical Trial.
Brief Title: The Erythropoietin NeuroProtective Effect: Assessment in CABG Surgery (TENPEAKS)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Calgary Health Region (Other); Ortho Biotech, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 17747
Record Dates: First submitted 2006-06-12; First posted 2006-06-13 (Estimated); Last update posted 2007-11-27 (Estimated); Status verified 2007-11

CONDITIONS: Cardiac Surgery; Brain Injury
Keywords: Cardiac bypass surgery
MeSH Terms: conditions — Brain Injuries

INTERVENTIONS:
Drug: Human recombinant erythropoietin

SUMMARY:
Context: Neurocognitive dysfunction complicates coronary artery bypass graft surgery. Neurocognitive dysfunction is a measurable problem with thinking. Erythropoietin may be a neuroprotectant.

Objective: To investigate the feasibility and safety of three doses of human recombinant erythropoietin to reduce neurocognitive dysfunction in coronary artery bypass graft patients.

DETAILED DESCRIPTION:
Coronary artery bypass surgery (CABG) is performed each year on over 500,000 patients in the US and almost 30,000 patients in Canada to treat coronary artery disease. However, it is complicated by a significant postoperative risk of neurologic sequelae, including stroke and neurocognitive dysfunction (NCD). Clinically overt stroke, which may be seen in 1-4% of patients, is far less common than NCD, which is reported in approximately 50-75% of patients at discharge, 20-50% at 6 weeks and up to 40% at five years.Human recombinant erythropoietin (rh-Epo) is not only approved in this population for prophylactic use to reduce blood transfusions, but has become an agent of intense interest for neuroprotection as a result of in vitro data, animal experiments, and now, two promising preliminary trials in human patients. There are not, however, any pilot data by which to estimate an appropriate dose or treatment effect of rh-Epo on NCD specifically. It is imperative both to refine estimates of control group incidence rates, treatment effect and test variability in CABG, as well to demonstrate the feasibility and safety of a study protocol, prior to embarking on a larger randomized controlled trial powered with an adequate sample size to investigate the efficacy of rh-Epo in the reduction of peri-operative NCD. We propose a six month prospective study in CABG patients to investigate the feasibility and safety of three prophylactic doses of human recombinant erythropoietin (rh-Epo) in a randomized, placebo controlled study. The four study arms are: placebo, 375 U/kg, 750 U/kg, or 1500 U/kg of human recombinant erythropoietin intravenously divided in three doses, the day before, the day of and the day after surgery. The primary outcomes of this pilot will be study feasibility and patient safety as measured by ICU and Hospital length of stay, 28 day all cause mortality, and incidence of morbidity including pure red cell aplasia (PRCA), stroke, myocardial infarction, re-operation, deep vein thrombosis, and pulmonary thromboembolism. The secondary outcome will be the incidence of neurocognitive dysfunction among the four study arms and between placebo and rh-Epo at any dose. As well, little is known about the pharmacology of rh-Epo in crossing the blood-brain barrier. In those patients receiving a spinal anesthetic in addition to a general anesthetic as part of their normal care, CSF will be analyzed for rh-Epo concentration, and then compared to drug dose and serum level.

ELIGIBILITY:
Inclusion Criteria:

* First time cardiac surgical patients
* Elective or urgent on pump coronary artery bypass grafting (CABG)
* Age 45-75
* Signed, informed consent

Exclusion Criteria:

* Emergent CABG less than 48 hours from presentation
* Symptomatic cerebrovascular disease
* Atrial fibrillation
* Congestive Heart Failure within 2 weeks of surgery
* Malignancy or pre-malignant state within 5 years
* Significant Kidney disease (creatinine >150 umol/L)
* Significant Liver disease (Bilirubin > 20 umol/L)
* Significant Lung Disease (FEV1< 1.5 L, pO2 <70 on room air, pCO2 >45)
* Psychiatric Illness requiring medication
* Alcohol Abuse
* Less than Grade 7 education or inability to read
* Allergy to Eprex, past history of pure red cell aplasia
* Anemia or untreated iron deficiency
* Pregnancy

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32
Dates: Start 2004-09; Study Completion 2005-05

PRIMARY OUTCOMES:
Safety
Feasibility

SECONDARY OUTCOMES:
Incidence of Neurocognitive Dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: David Zygun, MD, Principal Investigator — University of Calgary and Calgary Health Region
Locations (1):
- Foothills Hospital, Calgary, Alberta, Canada